CLINICAL TRIAL: NCT05740449
Title: International Proof of Concept Therapeutic Stratification Trial of Molecular Anomalies in Relapsed or Refractory HEMatological Malignancies in Children, Subprotocol A: Decitabine / Venetoclax and Navitoclax in Pediatric Patients With Relapsed or Refractory Hematological Malignancies
Brief Title: HEM-iSMART-A: Decitabine / Venetoclax and Navitoclax in Pediatric Patients With Relapsed or Refractory Hematological Malignancies
Acronym: HEM-iSMART A
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company stopped development and production of one of the IMP's.
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other); IBFM (Industry); Fight Kids Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-501865-29-00
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Lymphoblastic Lymphoma (Precursor B-Lymphoblastic Lymphoma/Leukaemia) Recurrent; Lymphoblastic Lymphoma (Precursor T-Lymphoblastic Lymphoma/Leukaemia) Recurrent; Lymphoblastic Lymphoma (Precursor B-Lymphoblastic Lymphoma/Leukaemia) Refractory; Lymphoblastic Lymphoma (Precursor T-Lymphoblastic Lymphoma/Leukaemia) Refractory
Keywords: Acute lymphoblastic leukemia; Lymphoblastic lymphoma; Epigentic approach; decitabine; navitoclax; venetoclax; Relapse; Refractory; Children; Adolescents; Young adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Recurrence; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Decitabine; venetoclax; navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sub-study A - Epigenetic approach (Experimental): Decitabine / Venetoclax and Navitoclax.
  Each cycle lasts 28 days.
  Cycle 1: Decitabine is given 10 mg/m2 intravenous, once a day on 5 consecutive days (Day 1 - 5), venetoclax 400 mg adult equivalent dose, once a day, Day 1 - Day 28 orally, with a ramp-up dose on day 1 and navitoclax once a day, Day 3 - 28 orally depending on the weight of the patient (dose level 1).
  Cycle 2: Decitabine is given 10 mg/m2 intravenous, once a day on 5 consecutive days (Day 1 - 5), venetoclax 400 mg adult equivalent dose, once a day, Day 1 - Day 28 orally and navitoclax once a day, Day 1 - 28 orally depending on the weight of the patient (dose level 1).
  Patients in dose level 2: will receive decitabine 20 mg/m2 intravenous once a day on 5 consecutive days (Day 1 - 5).
  Patients in dose level -1: will receive venetoclax 200 mg adult equivalent dose, once a day, Day 1 - Day 28 orally.
  All patients receive age adapted intrathecal chemnotherapy.
  Interventions: Drug: Decitabine; Drug: Venetoclax; Drug: Navitoclax; Drug: intrathecal chemotherapy

INTERVENTIONS:
Drug: Decitabine — intravenous
Drug: Venetoclax — oral
Drug: Navitoclax — oral
Drug: intrathecal chemotherapy — IT: Methotrexate +/- prednisone/hydrocortisone/cytarabine according to the degree of central nervous involvement

SUMMARY:
HEM-iSMART is a master protocol which investigates multiple investigational medicinal products in children, adolescents and young adults (AYA) with relapsed/refractory (R/R) ALL and LBL. Sub-protocol A is a phase I/II trial evaluating the safety and efficacy of Decitabine / Venetoclax and Navitoclax in children and AYA with R/R pediatric ALL/LBL

DETAILED DESCRIPTION:
HEM-iSMART is a master protocol with sub-protocols. The overarching objective is that introducing targeted therapy using a biomarker driven approach for treatment stratification may improve the outcome of children with R/R acute lymphoblastic leukemia (ALL) and lymphoblastic lymphoma (LBL) It is characterized by a shared framework that allows for the investigation of multiple IMPs and generate pivotal safety and efficacy evidence within the sub-protocols to establish and define the benefits and risks of new treatments for children with R/R leukemia.

Sub-protocol A within HEM-iSMART, is a phase I/II, multicenter, international, open-label clinical trial designed to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of decitabine, venetoclax and navitoclax in children, adolescents and young with R/R ALL and LBL. The epigenetic approach may improve outcome for patients whose tumor lack molecular alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 4 years and 18 years of age at the time of first diagnosis and less than 21 years at the time of inclusion. Children must have a body weight ≥ 20 kg.
2. Performance status: Karnofsky performance status (for patients >12 years of age) or Lansky Play score (for patients ≤12 years of age) ≥ 50% (Appendix I).
3. Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study specific screening procedures are conducted, according to local, regional or national guidelines.
4. For all oral medications patients must be able to comfortably swallow capsules (except for those for which an oral solution is available or dissolving of tablets is allowed based on investigator brochure (IB); nasogastric or gastrostomy feeding tube administration is allowed only if indicated).
5. Patients must have had advanced molecular profiling and flow-cytometric analysis of their recurrent or refractory disease at a time-point before the first inclusion into this trial (see section 9.1 of this protocol for detailed description of the molecular diagnostics required). Drug response profiling and methylation is highly recommended but not mandatory. Patients with advanced molecular profiling at diagnosis may be allowed to be included after discussion with the sponsor.
6. Adequate organ function:

   * RENAL AND HEPATIC FUNCTION (Assessed within 48 hours prior to C1D1) :

     * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) for age or calculated creatinine clearance as per the Schwartz formula or radioisotope glomerular filtration rate ≥ 60 mL/min/1.73 m2.
     * Direct bilirubin ≤ 2 x ULN (≤ 3.0 × ULN for patients with Gilbert's syndrome).
     * Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 5 x ULN; AST/serum glutamic oxaloacetic transaminase/SGOT ≤ 5 x ULN. Note: Patients with hepatic disfunction related to the underling disease can be eligible even if they do not fulfill the aforementioned values for hepatic transaminases. In these cases, patients need to be discussed with the sponsor to confirm the eligibility.
   * CARDIAC FUNCTION:

     * Shortening fraction (SF) >29% (>35% for children < 3 years) and/or left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography or MUGA.
     * Absence of QTcF prolongation (QTc prolongation is defined as >450 msec on baseline ECG, using the Friedericia correction), or other clinically significant ventricular or atrial arrhythmia.

Exclusion Criteria:

1. Pregnancy or positive pregnancy test (urine or serum) in females of childbearing potential. Pregnancy test must be performed within 7 days prior to C1D1.
2. Sexually active participants not willing to use highly effective contraceptive method (pearl index <1) as defined in CTFG HMA 2020 (Appendix II) during trial participation and until 6 months after end of antileukemic therapy.
3. Breast feeding.
4. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome) in case of oral IMPs.
5. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to the study drugs, or drugs chemically related to study treatment or excipients that contraindicate their participation, including conventional chemotherapeutics (i.e. cytarabine and cyclophosphamide when applicable, intrathecal agents) and corticoids.
6. Known active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
7. Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion.
8. Subjects unwilling or unable to comply with the study procedures.
9. Patients who have previously received decitabine can not participate.
10. Patients who have previously received venetoclax or navitoclax separately can be eligible for this sub-study.
11. Patients who have consumed grapefruit, grapefruit products, Seville oranges (Including marmalade containing Seville oranges) or starfruit within 72 hours prior to the first dose of study drug
12. Patients who have received strong and moderate CYP3A4 inhibitors/inducers within 7 days prior to the first dose of study drug (also see Appendix VI of the Master Protocol).
13. Current use of a prohibited medication or herbal preparation or requires any of these medications during the study. See Section 7, Appendix III and or details. In general, CYP3A4 inhibitors/Pgp inhibitors, moderate or strong inducers of CYP3A4 or drugs inducing QTc changes (prolongation of the QT interval or inducing Torsade de Points) are not permitted.
14. Unresolved toxicity greater than NCI CTCAE v 5.0 ≥ grade 2 from previous anti-cancer therapy, including major surgery, except those that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profile of the study treatment (e.g., alopecia and/or peripheral neuropathy related to platinum or vinca alkaloid based chemotherapy) (Common Terminology Criteria for Adverse Events (CTCAE) (cancer.gov).
15. Active acute graft versus host disease (GvHD) of any grade or chronic GvHD of grade 2 or higher. Patients receiving any agent to treat or prevent GvHD post bone marrow transplant are not eligible for this trial.
16. Received immunosuppression post allogenic HSCT within one moth of study entry.
17. Wash-out periods of prior medication:

    1. CHEMOTHERAPY: At least 7 days must have elapsed since the completion of cytotoxic therapy, with the exception of hydroxyurea, 6-mercaptopurine, oral methotrexate and steroids which are permitted up until 48 hours prior to initiating protocol therapy. Patients may have received intrathecal therapy (IT) at any time prior to study entry.
    2. RADIOTHERAPY: Radiotherapy (non-palliative) within 21 days prior to the first dose of drug. Palliative radiation in past 21 days is allowed.
    3. HEMATOPOIETIC STEM CELL TRANSPLANTATION:

       * Autologous HSCT within 2 months prior to the first study drug dose.
       * Allogeneic HSCT within 3 months prior to the first study drug dose.
    4. IMMUNOTHERAPY: At least 42 days must have elapsed after the completion of any type of immunotherapy other than monoclonal antibodies (e.g. CAR-T therapy)
    5. MONOCLONAL ANTIBODIES AND INVESTIGATIONAL DRUGS: At least 21 days or 5 times the half-life (whichever is shorter) from prior treatment with monoclonal antibodies or any investigational drug under investigation must have elapsed before the first study drug.
    6. SURGERY: Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) / Recommended phase 2 dose (RP2D) | 3 years
  Defined as the highest dose level tested at which 0/6 or 1/6 patients experiences dose limiting toxicities (DLT) during course 1 with at least 2 patients experiencing DLT at the next higher dose.
Phase II: Best overall response rate (ORR) | 6 years
  For patients with leukemia: CR and MRD response after 1 cycle of treatment. This includes determination of CR, CRp, CRi and minimal residual disease (MRD) negativity rate in patients suffering from overt morphological relapse of T-ALL at time of enrolment (morphological disease (M2/M3)), and the MRD negativity rate in those that entered with high-MRD levels but in morphological CR. These results will together be presented as a composite endpoint Overall Response rate (ORR). MRD negativity will be defined as ≤1x10-4 as generated by multi-parameter flow cytometry.
  For patients with lymphoma: Response in LBL patients is defined as CR, PR, minor response (MR) as defined in International pediatric NHL response criteria. In case of bone-marrow involvement MRD will be taken into account.

SECONDARY OUTCOMES:
Overall survival (OS) | 7 years
  Defined as time from C1D1 until death of any cause.
Event-free survival (EFS) | 7 years
  Defined as time from C1D1 to the first event (subsequent relapse after CR (including molecular reappearance), death of any cause, failure to achieve remission (CR, CRp or CRi), or secondary malignancy).
Cumulative incidence of relapse (CIR) | 7 years
  Estimate of the risk, that a patient will develop a relapse over a specified period of time.
Number of patients proceeding to hematopoietic stem cell transplantation (HSCT) after the experimental therapy. | 7 years
  The rate of those proceeding to subsequent allogenic HSCT
Cumulative overall response rate (ORR) | 7 years
  Defined as the CR, CRp, CRi and MRD negativity rates after more than 1 cycle of treatment
Rate of dose limiting toxicities (DLTs) | 7 years
  Number of participants with dose limiting toxicities (DLTs)
Peak plasma concentration (Cmax) | 6 years
  Estimation of decitabine, venetoclax and navitoclax Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Michel Zwaan, Prof. Dr., Study Chair — Princess Maxima Center for Pediatric Oncology; Andrej Lissat, MD, PhD, Principal Investigator — Charité
Locations (1):
- Princess Máxima Center for Pediatric Oncology, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be used to generate a publication
Supporting Information: CSR
Time Frame: CSRs will also be provided at the end of specific sub-protocols or specific phases of a sub-protocol, and when needed for regulatory purposes.
  Examples for generating 'primary CSRs' may include:
  After Last Patient Last Visit (LPLV) in a study having ORR as endpoint After the RP2D is determined in a Phase I part of a given sub-protocol After the follow-up of a specific sub-protocol is completed.
Access Criteria: A summary of the study results will be made public via clinicaltrials.gov as well as to Ethical committees/ Health Authorities and all participating patients by providing them through their treating physicians a patient letter with a summary of the results.